CLINICAL TRIAL: NCT02803294
Title: THE TORCH TRIAL：Transcatheter Aortic Valve Replacement Single Center Registry in Chinese Population
Brief Title: Transcatheter Aortic Valve Replacement Single Center Registry in Chinese Population
Acronym: TORCH
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Jian'an Wang,MD,PhD, President of Second Affiliated Hospital, School of Medicine, Zhejiang University & Chief of Cardiology, Second Affiliated Hospital, School of Medicine, Zhejiang University, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAHZJU CT006
Record Dates: First submitted 2016-06-07; First posted 2016-06-16 (Estimated); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Symptomatic Aortic Stenosis
MeSH Terms: interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aortic Stenosis/regurgitation (Experimental): Transcatheter aortic valve replacement
  Interventions: Procedure: transcatheter aortic valve replacement

INTERVENTIONS:
Procedure: transcatheter aortic valve replacement

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of transcatheter aortic valve replacement in Chinese population.

DETAILED DESCRIPTION:
Subjects enrolled are those who undergo physical exams and screening tests and were classified as a patient with symptomatic aortic stenosis or severe aortic regurgitation. They are then performed transcatheter aortic valve replacement.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic aortic stenosis/regurgitation
* Subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.
* The subject agrees to comply with specified follow-up evaluations and to return to the investigational site where the procedure was performed.
* Patients are technical and anatomical eligible for interventions

Exclusion Criteria:

* A known hypersensitivity or contraindication to any of the following which cannot be adequately pre-medicated: Aspirin Heparin (HIT/HITTS) and bivalirudin Nitinol (titanium or nickel) Ticlopidine and clopidogrel Contrast media
* Subject refuses a blood transfusion.
* Other medical, social, or psychological conditions that in the opinion of an Investigator precludes the subject from appropriate consent.
* Life expectancy is less than one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2016-06; Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Death from any cause | 1 year

SECONDARY OUTCOMES:
stroke | 30days, 6months,1 year,2 years, 3 years, 4 years, 5 years，10 years
death from cardiac causes | 30days, 6months,1 year,2 years, 3 years, 4 years, 5 years，10 years
myocardial infarction | 30days, 6months,1 year,2 years, 3 years, 4 years, 5 years，10 years
repeated hospitalization | 30days, 6months,1 year,2 years, 3 years, 4 years, 5 years， 10 years
acute kidney injury | 30days, 6months,1 year,2 years, 3 years, 4 years, 5 years，10 years
vascular complications | 30days, 6months,1 year,2 years, 3 years, 4 years, 5 years,10 years
bleeding events | 30days, 6months,1 year,2 years, 3 years, 4 years, 5 years，10 years
device success | 30days, 6months,1 year,2 years, 3 years, 4 years, 5 years，10 years
  Absence of procedural mortality and correct positioning of a single prosthetic valve into the proper anatomical location with intended performance of the prosthetic heart valve (no prosthesis-patient mismatch and mean aortic valve gradient <20 mmHg or peak velocity < 3 m/s, and no moderate or severe paravalvular regurgitation)
Functional Improvement from baseline per New York Heart Association functional classification | 30days, 6months,1 year,2 years, 3 years, 4 years, 5 years，10 years
permanent pacemaker implantation | 30days, 6months,1 year,2 years, 3 years, 4 years, 5 years，10 years
  number of patients who develop permanent third-degree or type 2(Mobitz) Secondary atrioventricular block after transcatheter aortic valve replacement and need permanent pacemaker implantation.
transcatheter valve failure | 30days, 6months,1 year,2 years, 3 years, 4 years, 5 years，10 years
  leaflet thrombosis formation, reduced leaflet motion or leaflet thickening of the prosthetic valve
changes in ascending aorta diameter | 1 year,2 years, 3 years, 4 years, 5 years，10 years
Death from all causes | 30 days, 6 months,1 year,2 years, 3 years, 4 years, 5 years，10 years

CONTACTS AND LOCATIONS:
Overall Officials: Jian-an Wang, MD,PhD, Principal Investigator — Second Affiliated Hospital of Zhejiang University School of Medicine
Locations (1):
- The Second Affiliated Hospital, School of Medicine at Zhejiang University, Hanzhou, Zhejiang, China

REFERENCES:
- [Derived] Fan J, Chen J, Zhu G, Xu Y, Ng S, Dai H, Zhou D, Yidilisi A, Qi X, Liu X, Wang J. Impact of repositioning on brain injury following transcatheter aortic valve replacement with a self-expanding valve. Sci Rep. 2024 Jul 30;14(1):17554. doi: 10.1038/s41598-024-67748-6. PMID 39080364
- [Derived] Zhou Q, Wen J, Zhu Q, Fan J, Guan X, Chen X, He Y, Guo Y, Jiang J, Ding X, Pu Z, Huang Z, Li C, Zhang M, Liu X, Xu X, Wang J. Long-term prosthetic-associated subclinical thrombotic events evaluation by cardiac CTA after transcatheter aortic valve implantation: incidence and outcomes. Insights Imaging. 2024 May 30;15(1):125. doi: 10.1186/s13244-024-01681-0. PMID 38816554
- [Derived] Hu P, Chen H, Wang LH, Jiang JB, Li JM, Tang MY, Guo YC, Zhu QF, Pu ZX, Lin XP, Ng S, Liu XB, Wang JA. Elevated N-terminal pro C-type natriuretic peptide is associated with mortality in patients undergoing transcatheter aortic valve replacement. BMC Cardiovasc Disord. 2022 Apr 12;22(1):164. doi: 10.1186/s12872-022-02615-8. PMID 35413789
- [Derived] Fan J, Fang X, Liu C, Zhu G, Hou CR, Jiang J, Lin X, Wang L, He Y, Zhu Q, Ng S, Chen Z, Hu H, Liu X, Wang J, Leon MB. Brain Injury After Transcatheter Replacement of Bicuspid Versus Tricuspid Aortic Valves. J Am Coll Cardiol. 2020 Dec 1;76(22):2579-2590. doi: 10.1016/j.jacc.2020.09.605. PMID 33243378